CLINICAL TRIAL: NCT02860988
Title: Responsible Fatherhood Opportunities for Reentry & Mobility
Acronym: ReFORM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mountain Comprehensive Care Center (Other)
Collaborators: University of Kentucky (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 90FO0007-01-00
Record Dates: First submitted 2016-08-02; First posted 2016-08-10 (Estimated); Results first posted 2021-04-30 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Healthy
Keywords: Fatherhood; Relationships; Employment; Criminal Justice

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MCCC Treatment (Experimental): Participants in this condition received newly-supported reentry services to enhance fatherhood and parenting for individuals with substance use issues. These services focus on responsible parenting, economic stability and mobility, and healthy marriage and relationships.
  Interventions: Behavioral: MCCC treatment
- MCCC Comparison (No Intervention): Participants in this condition did not receive reentry services related to responsible parenting, economic stability and mobility, or healthy marriage and relationships.

INTERVENTIONS:
Behavioral: MCCC treatment — Participants in this condition received newly-supported reentry services to enhance fatherhood and parenting for individuals with substance use issues. These services focus on responsible parenting, economic stability and mobility, and healthy marriage and relationships.
  Arms: MCCC Treatment

SUMMARY:
The purpose of this study is to determine differences among incarcerated or recently incarcerated fathers who receive targeted services and those who do not.

DETAILED DESCRIPTION:
Individuals with a criminal justice background (either incarcerated or on community supervision) and substance use issues will have the opportunity to enroll in services provided by the Mountain Comprehensive Care Center to focus on enhancing fatherhood and family situations.

The primary research questions focus on gauging the intervention's effectiveness in improving healthy relationship and responsible fatherhood outcomes. The intervention has several components targeting parenting skills, job training, relationship education, and case management/reentry support. Primary research questions include:

1. Compared to the counterfactual condition, what is the impact of the intervention on parenting and co-parenting skills/behaviors, as measured by parental role satisfaction and confidence in parenting skills six months after release from incarceration?
2. Compared to the counterfactual condition, what is the impact of the intervention on the likelihood that the participant will be employed six months after release from incarceration?
3. Compared to the counterfactual condition, what is the impact of the intervention on the likelihood that the participant will be in a relationship six months after release from incarceration?

ELIGIBILITY:
Inclusion Criteria:

* Male inmates at specific eastern Kentucky jail sites who are at least 18 years of age and not previously screened for the study
* Participants for the local evaluation will be identified as eligible fathers who have been tried and convicted as an adult; within 3 to 9 months of release; are low-income; and may be an expectant father, a biological father, an adoptive father or a stepfather or who a person who is acknowledged as a father figure (e.g., grandfather) of a dependent child or young adult child up to 24 years of age, and interested in participation.

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were eligible if they were tried and convicted as adults; and were expectant or current adult fathers, including adoptive or step-fathers, or others acknowledged as a father figure of a dependent child or young adult up to 20 years of age.
Pre-assignment Details: Of the 704 screened, 248 (43%) did not meet eligibility criteria. Of those screened, 401 (57%) met eligibility criteria and all of those eligible completed a baseline survey (N=401).
Period: Overall Study
Arm/Group | MCCC Treatment | MCCC Comparison
Started | 201 | 200
Completed | 117 | 94
Not Completed | 84 | 106

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MCCC Treatment | MCCC Comparison | Total
Number analyzed (Participants) | 201 | 200 | 401
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 201 | 200 | 401
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.1 (9.0) | 36.9 (8.5) | 37.4 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 201 | 200 | 401
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 155 | 159 | 314
  Black or African American | 2 | 8 | 10
  More than one race | 1 | 1 | 2
  Unknown or not reported | 43 | 32 | 75
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 201 | 200 | 401
Age at time of first arrrest [Mean (Standard Deviation); unit: years] | 19.5 (6.9) | 18.7 (5.4) | 19.1 (6.2)
Number of arrests in lifetime [Mean (Standard Deviation); unit: arrests] | 22.9 (28.2) | 23.2 (33.8) | 23.1 (31.1)

OUTCOME MEASURES:

1. Primary Outcome: Parental Role Satisfaction
Description: A scale calculated by summing three times measuring happiness, closeness, and comforting interactions with the child. Total score range is 3-12, with higher scores indicating greater satisfaction.
Time Frame: 6-month follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MCCC Treatment | MCCC Comparison
Number analyzed (Participants) | 33 | 43
units on a scale | 11.9 (0.2) | 11.4 (1.6)
Statistical Analysis 1: Comparison: MCCC Treatment vs MCCC Comparison; Test type: Other — Two-sided tests versus a margin; p = 0.29, Regression, Linear — A priori threshold for statistical significance was set at 0.05; Mean Difference (Net) = 0.6

2. Primary Outcome: Number of Participants Employed
Description: The outcome is a dichotomous indicator of whether the participant currently has a job.
Time Frame: 6-month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | MCCC Treatment | MCCC Comparison
Number analyzed (Participants) | 117 | 94
Participants | 26 | 20
Statistical Analysis 1: Comparison: MCCC Treatment vs MCCC Comparison; Test type: Other — Two-sided tests versus a margin; p = 0.88, Regression, Logistic — A priori threshold for statistical significance was set at 0.05; Risk Difference (RD) = 0.9

3. Primary Outcome: Number of Participants in a Relationship
Description: The outcome measure is a dichotomous indicator of whether the participant is currently in a relationship.
Time Frame: 6-month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | MCCC Treatment | MCCC Comparison
Number analyzed (Participants) | 117 | 94
Participants | 47 | 37
Statistical Analysis 1: Comparison: MCCC Treatment vs MCCC Comparison; Test type: Other — Two-sided tests versus a margin; p = 0.89, Regression, Logistic — A priori threshold for statistical significance was set at 0.05; Risk Difference (RD) = 0.96

4. Secondary Outcome: Number of Participants With Recent In-person Contact With Child(Ren)
Description: The measure is a dichotomous indicator of whether the participant has seen their child in person during the past month.
Time Frame: 6-month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | MCCC Treatment | MCCC Comparison
Number analyzed (Participants) | 117 | 94
Participants | 58 | 50
Statistical Analysis 1: Comparison: MCCC Treatment vs MCCC Comparison; Test type: Other — Two-sided tests versus a margin; p = 0.61, Regression, Logistic — A priori threshold for statistical significance was set at 0.05; Risk Difference (RD) = -4.26

5. Secondary Outcome: Number of Participants With Recent Other Contact With Child(Ren)
Description: The measure is a dichotomous indicator of whether the participant has spoken with their child on the phone or sent their child letters within the past month.
Time Frame: 6-month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | MCCC Treatment | MCCC Comparison
Number analyzed (Participants) | 117 | 94
Participants | 69 | 52
Statistical Analysis 1: Comparison: MCCC Treatment vs MCCC Comparison; Test type: Other — Two-sided tests versus a margin; p = 0.67, Regression, Logistic — A priori threshold for statistical significance was set at 0.05; Risk Difference (RD) = 3.61

6. Secondary Outcome: Number of Participants That Participated in an Education or Job Training Program in the Past 30 Days
Description: The measure is a dichotomous indicator of whether the participant has participated in education or job training programs within the past month.
Time Frame: 6-month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | MCCC Treatment | MCCC Comparison
Number analyzed (Participants) | 117 | 94
Participants | 10 | 3
Statistical Analysis 1: Comparison: MCCC Treatment vs MCCC Comparison; Test type: Other — Two-sided tests versus a margin; p = 0.14, Regression, Logistic — A priori threshold for statistical significance was set at 0.05; Risk Difference (RD) = 5.23

7. Secondary Outcome: Partner Conflict Resolution
Description: The measure is a Likert-type (very/somewhat/not at all satisfied) response to whether the participant is satisfied with the way that they and their partner/spouse handle conflict. Total scores range 1-3, with higher scores indicating a greater level of satisfaction.
Time Frame: 6-month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MCCC Treatment | MCCC Comparison
Number analyzed (Participants) | 117 | 94
score on a scale | 1.4 (0.5) | 1.4 (0.5)
Statistical Analysis 1: Comparison: MCCC Treatment vs MCCC Comparison; Test type: Other — Two-sided tests versus a margin; p = 0.81, Regression, Linear — A priori threshold for statistical significance was set at 0.05; Mean Difference (Net) = 0.03

8. Secondary Outcome: Mental Health Distress
Description: The outcome measure is a scale calculated from six items measuring symptoms of anxiety and depression experienced in the past month. Total scores range from 6-30,w with higher scores indicating more frequent experience with symptoms (i.e., greater distress).
Time Frame: 6-month follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MCCC Treatment | MCCC Comparison
Number analyzed (Participants) | 117 | 94
units on a scale | 11.9 (5.8) | 11.2 (6.3)
Statistical Analysis 1: Comparison: MCCC Treatment vs MCCC Comparison; Test type: Other — Two-sided tests versus a margin; p = 0.74, Regression, Linear — A priori threshold for statistical significance was set at 0.05; Mean Difference (Net) = 0.31

ADVERSE EVENTS:
Time Frame: 6 months post-study enrollment
Arm/Group | MCCC Treatment | MCCC Comparison
All-Cause Mortality (participants affected / at risk) | 0/201 | 0/200
Serious Adverse Events (participants affected / at risk) | 0/201 | 0/200
Other Adverse Events (participants affected / at risk) | 0/201 | 0/200

LIMITATIONS AND CAVEATS:
The follow-up sample size (n=211; 53% follow-up) may have limited the ability to detect intervention effects. In addition, other measures than those used in this evaluation may have been more sensitive to differences between the intervention and counterfactual groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-09-29): https://cdn.clinicaltrials.gov/large-docs/88/NCT02860988/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-15): https://cdn.clinicaltrials.gov/large-docs/88/NCT02860988/SAP_001.pdf
  • Informed Consent Form (2020-09-29): https://cdn.clinicaltrials.gov/large-docs/88/NCT02860988/ICF_002.pdf